CLINICAL TRIAL: NCT02125435
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of ASP2408 Following Single Intravenous Doses in Healthy Subjects
Brief Title: A Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of ASP2408 Following Single Intravenous Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2408-CL-0101
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP2408
Keywords: Healthy subjects; ASP2408; pharmacokinetics
MeSH Terms: interventions — ASP2408

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP2408 dose escalation cohort (Experimental)
  Interventions: Drug: ASP2408
- Placebo dose escalation cohort (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP2408 — intravenous
  Arms: ASP2408 dose escalation cohort
Drug: Placebo — intravenous
  Arms: Placebo dose escalation cohort

SUMMARY:
The objective of this study is to assess the safety, tolerability, and pharmacokinetics (PK) of single ascending intravenous (IV) doses of ASP2408 in non-elderly, healthy male and female subjects and to evaluate the pharmacodynamics of ASP2408.

DETAILED DESCRIPTION:
This is single-dose escalation study composed of 8 sequential cohorts of healthy subjects receiving increasing doses of intravenously administered ASP2408 or matching placebo. Subjects will be confined in the clinic for 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject weighs at least 50 kg, and has a body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive.
* Results of subject's 12-lead electrocardiogram (ECG) are normal or, if abnormal, the abnormality is not clinically significant as determined by the investigator.
* Female subject must be at least two years postmenopausal OR surgically sterile (with documentation provided by a healthcare professional) and not pregnant or lactating.
* Male subject agrees to the use of male condoms until the end of study or 60 days post dose, whichever is longer.
* Subject is highly likely to comply with the protocol and complete the study.

Exclusion Criteria:

* Subject has a history of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy excluding adequately treated non-melanoma skin cancer.
* Subject has a history of severe allergic or anaphylactic reactions.
* Subject is a female of child-bearing potential.
* Subject has a history of consuming more than 14 units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/ substance abuse within past 2 years (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits).
* Subject has a positive test for alcohol or drugs of abuse.
* Subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic check-in.
* Subject has a past history of opportunistic infection.
* Subject has a supine mean systolic blood pressure < 90 or > 160 mmHg and a mean diastolic blood pressure < 50 or > 90 mmHg, or mean pulse rate higher than 100 beats per min (bpm).
* Subject is known positive for human immunodeficiency virus (HIV) antibody.
* Subject has a positive TB skin test or Quantiferon Gold test or T-SPOT® test at Screening.
* Subject has a positive test for hepatitis C antibody, or positive test for hepatitis B surface antigen (HBsAg), or positive hepatitis B core antibody.
* Subject's laboratory test results:

  * alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), are greater than 1.5 times the upper limit of normal
  * are outside the normal limits and considered by the investigator to be clinically significant with regard to the remaining per-protocol laboratory tests.
* Subject received any vaccine within 60 days prior to study drug administration.
* Subject received any systemic immunosuppressant agent within 2 months prior to study drug administration.
* Subject has previously received any antibody or therapeutic biologic product prior to study drug administration.
* Subject received any systemic steroid within 2 months or steroid inhaler within 1 month prior to study drug administration.
* Subject has had treatment with prescription, non-prescription or complementary and alternative medicines (CAM) within 14 days prior to study drug administration.
* Subject has received an experimental agent within 30 days or five half-lives, whichever is longer, prior to study drug administration.
* Subject is participating in another clinical trial or has participated in another dose group of the current trial.
* Subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on Day -1.
* Subject has a history of heavy smoking or has used tobacco-containing products and nicotine or nicotine-containing products in the past six months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of ASP2408:AUClast | Days 1-8, 15, 22, 29, 43, 60, 90
  Area Under the Concentration - Time curve from time 0 up to the last quantifiable concentration (AUClast)
Pharmacokinetic parameter of ASP2408: AUCinf | Days 1 -8, 15, 22, 29, 43, 60, 90
  Area Under the Concentration - Time curve from time 0 extrapolated to infinity (AUCinf)
Pharmacokinetic parameter of ASP2408:Cmax | Days 1-8, 15, 22, 29, 43, 60, 90
  Maximum concentration (Cmax)
Safety assessed by adverse events, laboratory tests, immunoglobulin, 12-lead electrocardiograms (ECGs), vital signs and anti-2408 antibody formulation | up to 90 days

SECONDARY OUTCOMES:
Composite of pharmacokinetics of ASP2408: tmax, t1/2, Vz, CLtot | Days 1-8, 15, 22, 29, 43, 60, 90
  Time to attain Cmax (tmax), apparent terminal elimination half-life (t1/2), Terminal phase volume (Vz), Total Body Clearance (CLtot)
Pharmacodynamic parameters of ASP2408: CD80 and CD86 receptor occupancy | Days 1-3, 5, 8, 15, 22, 29, 43, 60, 90
Total lymphocyte count | Days 1-3, 5, 8, 15, 22, 29, 43, 60, 90
Peripheral lymphocyte subset quantification | Days 1-3, 5, 8, 15, 22, 29, 43, 60, 90

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- PAREXEL International, Baltimore, Maryland, United States